CLINICAL TRIAL: NCT00589524
Title: Comparison of Non-invasive Coronary CT With IVUS for the Detection of Coronary Artery Vasculopathy in a Cardiac Transplant Population
Brief Title: Comparison of Coronary CT With IVUS in Heart Transplant Population
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficult recruitment -
Sponsor: Mayo Clinic (Other)
Responsible Party: Amir Lerman, M.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 06-007193
Record Dates: First submitted 2007-12-21; First posted 2008-01-09 (Estimated); Last update posted 2012-01-16 (Estimated); Status verified 2012-01

CONDITIONS: Heart Transplantation
Keywords: blocked arteries; narrowing arteries; IVUS; CT
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Computed tomography (CT) — Computed tomography (CT), as performed by Dual Source Computed Tomography (DSCT)(Siemens Medical Solutions Germany) to be conducted no sooner than 3 days before or after cardiac catheterization, but with 3 months of the cardiac cath.
  Other Names: DSCT Scanner, 4D scanner serial number 60011

SUMMARY:
To compare results of Intravascular Ultrasound (which occurs during cardiac catheterization) with Computed Tomography (CT) scan to detect blockages or narrowing of the arteries that feed the heart. These will be studied in the cardiac transplant population.

ELIGIBILITY:
Inclusion Criteria:

* Heart transplant patients coming to the Cardiac Cath Lab for their yearly angiogram which includes intravascular ultrasound (IVUS)

Exclusion Criteria:

* Patients with a history of allergic reactions to contrast material Creatine >1.5 Clinical or hemodynamic instability Those who are unable to consent for enrollment into the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
To determine if Computed Tomography (CT) of the arteries that feed the heart is more sensitive than Intravascular Ultrasound (IVUS) which is performed during cardiac catheterization | within 3 months of cardiac cath with IVUS

CONTACTS AND LOCATIONS:
Overall Officials: Amir Lerman, MD, Principal Investigator — Mayo Clinic